CLINICAL TRIAL: NCT01906164
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 3-Part Study of Orally Administered ALS-008176 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Dosing, Multiple Ascending Dosing and Food-effect in Healthy Volunteers
Brief Title: Study of Single and Multiple Doses of ALS-008176 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALS-8176-501; 2012-004894-14 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-07-24 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- ALS-008176 (Experimental)
  Interventions: Drug: ALS-008176
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALS-008176
  Arms: ALS-008176
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics (PK) of orally administered ALS-008176 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18-55 years of age, in good health with screening laboratory values within limits specified by the protocol
* Body mass index 18-30 kg/m2
* Female subjects must be of non-childbearing potential; male subjects must be surgically sterile or practicing birth control

Exclusion Criteria:

* Clinically significant or uncontrolled medical illness
* Use, or anticipated use during conduct of the study, of concomitant medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
Safety data including, but not limited to, tabulation of adverse events, physical exams, vital signs, 12-lead ECGs and clinical lab results (including chemistry, hematology, and urine) | 11 days

SECONDARY OUTCOMES:
PK parameters of ALS-008176 and metabolites in plasma following single dose administration: Cmax, tmax, t1/2, CL/F and Vdss/F (not for metabolites), AUC0-24h, AUC0-inf or AUC0-last | 11 days
PK parameters of ALS-008176 and metabolites in plasma following repeat dose administration: Cmax, Cmin, tmax, t1/2, CL/F and Vdss/F (not for metabolites), AUC0-24h , AUC0-last and AUC0 tau | 11 days
Urinary excretion and concentrations of ALS-008176 and metabolites after a single oral dose and multiple doses in healthy volunteers in fasted conditions | 11 days
PK parameters of ALS-008176 and metabolites in plasma after a single oral dose in healthy volunteers in fasted conditions as compared with fed conditions: Cmax, tmax, t1/2, CL/F and Vdss/F (not for metabolites), AUC0-24h, AUC0-inf or AUC0-last | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McClure, M.D., Study Director — Alios BioPharma
Locations (1):
- Investigational Site, Rennes, France